CLINICAL TRIAL: NCT01137084
Title: Liver Transplantation Results in Hepatocellular Carcinoma Patients With Immunosuppression Without Steroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other); Nanchang University (Other); Zhejiang University (Other); Shanghai Changzheng Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20100603
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Immunosuppression; Hepatocellular Carcinoma; Liver Transplantation; Post-operative Complications
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- a steroid immunosuppression protocol (Active Comparator)
  Interventions: Drug: solu medrol
- a steroid-free immunosuppression protocol (Active Comparator): without steroid
  Interventions: Drug: a steroid-free immunosuppression protocol

INTERVENTIONS:
Drug: solu medrol — total dose 20mg/kg, including first dose 10mg/kg, rest of drug given within one weeks after liver transplantation
  Arms: a steroid immunosuppression protocol
Drug: a steroid-free immunosuppression protocol — receive immunosuppression with Basiliximab(20mg/day,twice following transplantation) and tacrolimus(0.06/kg/d,twice a day) without steroids.
  Arms: a steroid-free immunosuppression protocol

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of a steroid-free immunosuppression protocol in Hepatocellular Carcinoma (HCC) patients.

ELIGIBILITY:
Inclusion Criteria:

* All liver transplantation patients with hepatocellular carcinoma in our center between Jan 2005 and Dec 2009 were potentially eligible for enrollment

Exclusion Criteria:

* the recipient pass away within 3 month following up liver transplantation
* Inability to provide written informed consent prior to study entry
* acute rejection are treated only with steroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
patient and graft survival | Over 12-month after liver transplantation
  patient and graft survival include surviral rate and recurrence-free survival rate

SECONDARY OUTCOMES:
Postoperative complications | Over 12-month after liver transplantation
  Postoperative complications include acute rejection, infection, metabolic complications and hepatitis B-virus recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Hai Peng, MD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Foroncewicz B, Mucha K, Ryszkowska E, Ciszek M, Ziolkowski J, Porowski D, Krawczyk M, Paczek L. Safety and efficacy of steroid-free immunosuppression with tacrolimus and daclizumab in liver transplant recipients: 6-year follow-up in a single center. Transplant Proc. 2009 Oct;41(8):3103-6. doi: 10.1016/j.transproceed.2009.07.082. PMID 19857686
- [Result] Sutherland S, Li L, Concepcion W, Salvatierra O, Sarwal MM. Steroid-free immunosuppression in pediatric renal transplantation: rationale for and [corrected] outcomes following conversion to steroid based therapy. Transplantation. 2009 Jun 15;87(11):1744-8. doi: 10.1097/TP.0b013e3181a5df60. PMID 19502970
- [Result] Li L, Chang A, Naesens M, Kambham N, Waskerwitz J, Martin J, Wong C, Alexander S, Grimm P, Concepcion W, Salvatierra O, Sarwal MM. Steroid-free immunosuppression since 1999: 129 pediatric renal transplants with sustained graft and patient benefits. Am J Transplant. 2009 Jun;9(6):1362-72. doi: 10.1111/j.1600-6143.2009.02640.x. Epub 2009 May 13. PMID 19459814
- [Result] Mastrobuoni S, Ubilla M, Cordero A, Herreros J, Rabago G. Two-dose daclizumab, tacrolimus, mycophenolate mofetil, and steroid-free regimen in de novo cardiac transplant recipients: early experience. Transplant Proc. 2007 Sep;39(7):2163-6. doi: 10.1016/j.transproceed.2007.06.073. PMID 17889125
- [Result] Humar A, Crotteau S, Gruessner A, Kandaswamy R, Gruessner R, Payne W, Lake J. Steroid minimization in liver transplant recipients: impact on hepatitis C recurrence and post-transplant diabetes. Clin Transplant. 2007 Jul-Aug;21(4):526-31. doi: 10.1111/j.1399-0012.2007.00683.x. PMID 17645714